CLINICAL TRIAL: NCT05141071
Title: Effect of Ivabradine on Microcirculation and Cardiac Output in Patients Diagnosed With Septic Shock (Open-label Randomized Controlled Study)
Brief Title: Effect of Ivabradine on Microcirculation and Cardiac Output in Septic Shock Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amr Kamal Zahran, Lecturer of Anesthesia and Intensive care medicine, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MD-214 -2019
Record Dates: First submitted 2021-08-12; First posted 2021-12-02 (Actual); Last update posted 2022-09-01 (Actual); Status verified 2022-08

CONDITIONS: Septic Shock
Keywords: Micro-circulation; Septic shock; Cardiac output; Ivabradine
MeSH Terms: conditions — Shock, Septic | interventions — Ivabradine; Saline Solution

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ivabradine (Experimental): In the study group, Ivabradine(I) group; patients will receive an enteral Ivabradine (dissolved in distilled water) 5mg twice daily (every 12 hours) via a naso-gastric tube.
  Interventions: Drug: Ivabradine 5mg Tab
- Placebo (Placebo Comparator): the control group, Placebo (P) group; patients will receive 50 ml of saline twice daily also via a naso-gastric tube.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ivabradine 5mg Tab — Ivabradine will be administrated enterally
  Other Names: procoralan, ATC code: C01EB17
  Arms: Ivabradine
Drug: Placebo — 50 ml of saline will be administrated enterally
  Other Names: 0.9% saline solution
  Arms: Placebo

SUMMARY:
Persistent tachycardia in sepsis or multi-organ dysfunction syndrome (MODS) is an ominous sign. This usually comes under control with judicious use of antibiotics, fluid resuscitation, sedation. Uncontrolled tachycardia in systemic inflammatory response syndrome and sepsis deprives the heart muscle of oxygen. As it progresses, insufficient heart muscle nutrition eventually leads to myocardial dysfunction. It can also present as heart failure. In acute coronary syndromes, beta blockers are used to control heart rate. However in MODS, it cannot be used due to hemodynamic instability and worsened myocardial function.

Sinoatrial (SA) myocytes are the pacemaker cells in the heart. Pacemaker activity involves several ionic currents that influences spontaneous depolarization of SA node including I(f) current. The word I(f) means funny, because this current has unusual properties as compared with other currents known at the time of its discovery. It is one of the most important ionic current for regulating pacemaker activity in SA node.

Ivabradine is an I(f) current inhibitor in SA node. Currently, it is the only agent shown to clinically lower heart rate with no negative inotropism or effects on conduction and contractility.so usage of Ivabradine to control tachycardia in patients with septic shock may help to improve myocardial filling and cardiac output.

Marcos L.Miranda et al. found that Ivabradine was effective in reducing microvascular derangements evoked by experimental sepsis, which was accompanied by less organ dysfunction. These results suggest that ivabradine yields beneficial effects on the microcirculation of septic animals.

No data found on effect of Ivabradine on the microcirculation of human. In this study the investigators will investigate the effect of Ivabradine on perfusion in capillary circulation using Cytocam video microscope, Braedius®.

DETAILED DESCRIPTION:
All patients will be monitored with non-invasive arterial blood pressure, five-lead electrocardiography (ECG), pulse oximetry, and invasive arterial pressure (AP) obtained from a radial arterial catheter.

Upon ICU admission, according to the investigators' institutional protocol, fluid responsiveness will be done for all enrolled patients to determine the need for fluid therapy (fluid responsiveness is defined as an increase in the stroke volume (SV) by 15% after infusing 500 ml crystalloids). Fluid boluses will be repeated till the patients become fluid unresponsiveness. If mean arterial pressure (MAP) remained < 65 mm Hg after administration of the initial fluid bolus, norepinephrine infusion will be titrated to maintain MAP ≥ 65 mmHg.

After establishment of blood pressure and normovolemia, the patient will receive either placebo or Ivabradine according to the group randomization.

Assessment of microcirculation:

Sublingual microcirculatory measurements will be performed with an incident dark-field illumination device Cytocam- incident dark-field illumination (IDF), Braedius Medical, Huizen, Netherlands). The new technology Cytocam-IDF imaging device consists of a pen-like probe incorporating IDF illumination with a set of high-resolution lenses projecting images on to a computer-controlled image sensor synchronized with a short-pulsed illumination light. Flow characteristics of the microvasculature will be quantified using the microvascular ﬂow index (MFI), a semiquantitative technique consistent with recommendations from a consensus conference on microcirculatory image analysis in human subjects.The image is divided into four quadrants and the vessels <20 μ m diameter are assigned a score based on the predominant flow characteristics of the vessels in that quadrant (0 = absent flow; 1 = intermittent; 2 = sluggish; 3 = normal). The values in each quadrant will be averaged to give an MFI for each sublingual site at each time point. To determine heterogeneity of perfusion, the flow heterogeneity index will be calculated as the highest MFI minus the lowest MFI divided by the mean MFI. A quantitative measurement of the total vessel density (TVD), perfused vessel density (PVD), and proportion of perfused vessels (PPV), will also be taken automatically with dedicated software (Cytocam video microscope, Braedius®, Netherlands). The observer will be well-trained and experienced with offline analysis. On all videos, post-process contrast enhancement will be applied. Thereafter videos will be blinded and anonymized so that the observer will not be aware of the used drug.

Assessment of cardiac output using LiDCOrapid Examination:

A 20-G arterial catheter will be placed in the radial artery and connected to the standard monitor. LiDCOrapid (LiDCO Ltd, Cambridge, UK) will be connected to the monitor and data will be extracted from the AP line. Values for AP and heart rate extracted by LiDCOrapid will be in all patients within 5% of the standard monitor's displayed values (datex monitor). The LiDCO system is based on a PulseCO algorithm for calculating nominal cardiac output (CO), SV and heart rate from AP waveform characteristics.

Assessment of metabolic parameters:

Metabolic parameters including central venous saturation (ScvO2), central venous-arterial blood carbon dioxide partial pressure difference (Pv-aCO2), and arterial lactate will be recorded. Simultaneous blood gas measurements will be obtained from arterial and central venous catheters. Blood gas analysis will be performed and arterial lactate concentration will be determined using the GEM Premier 3000 (Instrumentation Laboratory, Bedford, MA, USA). ScvO2 will be calculated from a sample taken from the central venous catheter, the tip of which will be confirmed to be in the superior vena cava near or at the right atrium by radiography. The (Pv-aCO2) will be calculated as the difference between the partial pressures of central venous carbon dioxide (PcvCO2) and arterial carbon dioxide (PaCO2).

ELIGIBILITY:
Inclusion criteria:

* Age > 18 years.
* Patients admitted to ICU with septic shock.

Exclusion criteria:

* Patients contraindicated to begin oral feeding (NPO patients).
* Patients diagnosed with arrhythmia.
* Patients taking drugs with known or suspected interactions with ivabradine (strong CYP3A4 inhibitors and QT-prolonging agents) within five half-lives prior to inclusion and during the first 24 h of the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2021-11-25 (Actual); Primary Completion 2022-05-25 (Actual); Study Completion 2022-06-05 (Actual)

PRIMARY OUTCOMES:
Microvascular ﬂow index | 6 hours after administration of Ivabradine or Placebo.
  absent (0), intermittent (1), sluggish (2), or normal (3)

SECONDARY OUTCOMES:
Microvascular ﬂow index | Before drug administration and at 1, 12, and 24 hours thereafter.
  absent (0), intermittent (1), sluggish (2), or normal (3)
Total vessel density | Before drug administration and at 1, 6,12, and 24 hours thereafter.
  mm/mm2
Percentage of perfused vessels | Before drug administration and at 1, 6,12, and 24 hours thereafter.
  Percentage
Cardiac output | Before drug administration and at 1, 6,12, and 24 hours thereafter.
  litres per minute
Heart rate | Before drug administration and at 1, 6,12, and 24 hours thereafter.
  beats per minute
Central venous saturation | Before drug administration and at 1, 6,12, and 24 hours thereafter.
  Percentage
Central venous-arterial blood carbon dioxide partial pressure difference | Before drug administration and at 1, 6,12, and 24 hours thereafter.
  mmHg
Mean arterial blood pressure | Before drug administration and at 1, 6,12, and 24 hours thereafter.
  mmHg
ICU length of stay | from the date of patient recruitment till the date of discharge from the ICU or the date of death, assessed up to 28 days
  Days
28 days ICU mortality | 28 days after ICU admission
  Percentage

CONTACTS AND LOCATIONS:
Overall Officials: Amr K Abdelhakim, MD, Principal Investigator — Cairo University
Locations (1):
- Kasr Alainy Hospital, Cairo, Manial, Egypt